CLINICAL TRIAL: NCT06284577
Title: Probiotic Supplementation, Quality of Life and Gut Health in Pediatric Patients With Cystic Fibrosis
Brief Title: Quality of Life and Gut Health in Pediatric Patients With Cystic Fibrosis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: Norwegian National Advisory Unit on Rare Disorders, Oslo University Hospital (Unknown)
Responsible Party: Principal Investigator, Magnhild L. P. Kolsgaard, Dietitian, PhD, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 677186
Record Dates: First submitted 2024-02-12; First posted 2024-02-29 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Cystic Fibrosis in Children
Keywords: Cystic Fibrosis; Children; Microbiota; Quality of life; Probiotic supplement; CFTR modulators; elexacaftor-tezacaftor-ivacaftor
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotics (Experimental): Participants will recieve a multi-strain probiotic daily for 6 months
  Interventions: Dietary Supplement: Multistrain Probiotic
- Placebo (Sham Comparator): Participants will recieve maltodextrin daily for 6 months
  Interventions: Dietary Supplement: Placebo - maltodextrin

INTERVENTIONS:
Dietary Supplement: Multistrain Probiotic — Participants will recieve a multi-strain probiotic daily for 6 months
  Arms: Probiotics
Dietary Supplement: Placebo - maltodextrin — Participants will recieve placebo/ maltodextri daily for 6 months
  Arms: Placebo

SUMMARY:
The aim of the present study is to investigate the effect of probiotic supplementation on GI related quality of life, through a randomised placebo-controlled clinical trial. Moreover, the invetigators wish to study CF microbiota and intestinal inflammation in the setting of probiotic supplementation and newly started treatment with a highly effective CF-specific treatment, elexacaftor-tezacaftor-ivacaftor (ETI). The proposed project has the potential to increase QoL and decrease GI morbidity in children with CF. If successful, the results of this study can contribute to alter the care of CF patients by including supplementation of probiotics in routine CF care. Morever, the study can provide much needed insights to GI microbiota and inflammation in pediatric CF patients.

DETAILED DESCRIPTION:
The project targets pediatric patients with cystic fibrosis (CF), and has to work packages (WP). WP1 is an observational study, and WP2 is a randomised placebo-controlled clinical trial. The goal of the study is to investigate the effect of probiotics on pediatric CF patients' quality of life (QoL). Moreover the investigators wish to explore effects of both a highly effective CFTR modulator and probiotics on gut microbiota and intestinal inflammation.

The primary question it aims to answer are:

• Can probiotics improve GI related QoL in children with CF?

Secondary aims are to:

* Investigate GI microbiota and GI inflammation before and after commencement of the highly effective triple-combination elexacaftor-tezacaftor-ivacaftor (ETI)
* Explore GI microbiota before and after treatment with probiotics vs. placebo
* Study intestinal inflammation before and after treatment with probiotics vs. placebo
* Examine body composition and its relation to lung function

In WP1 participants will during routine examination before starting treatment with ETI be asked to deliver stool samples, and fill in QoL questionnaires. In WP2 participants will be randomized to intervention with probiotics or placebo, and the same parameters as in WP1 will also be collected.

ELIGIBILITY:
Inclusion criteria for WP1:

* CFTR mutations eligible for treatment with ETI
* Age 2-18 years. Majority of patients will be 2-6 years of age as ETI was approved from 6 years of age in 2022, and will be available for children above 2 years from 2024.
* Included in the Norwegian CF Register and consented to participation in CF general research biobank

Exclusion criteria for WP1:

* Other CFTR modulators commenced the last 6 months before inclusion
* Use of probiotics or prebiotics last 2 months
* Current pulmonary exacerbation

Inclusion criteria for WP2:

* Age 3-18 years
* CFTR modulator treatment naïve or treated with CFTR modulator for at least 6 months
* Included in the Norwegian CF Register and consented to participation in CF general research biobank

Exclusion criteria for WP2:

* CFTR modulators commenced the last 6 months before inclusion
* Use of probiotics or prebiotics last 2 months
* Current pulmonary exacerbation

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-01-02 (Actual); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Changes in GI related QoL using the questionnaire PedsQL GI | 0-6 months
  PEDsQL GI has been validated for use in the CF population. Participants will be scored before and 6 months after treatment start with ETI (WP2), and before and after 6 months treatment with probiotics vs placebo (WP2).

SECONDARY OUTCOMES:
Changes in microbiota | 0-6 months
  Stool samples for microbiota will be collected using a collection kit provided to the participants at recruitment, and then after 6 month of ETI treamtment (WP1), or probiotic/placebo (WP2). Microbiota analysis will be done using 16s rRNA amplicon sequencing and reduced metagenome sequencing.
Changes in intestinal inflammation | 0-6 months
  Stool samples for gut inflammation markers will be collected using a collection kit provided to the participants at recruitment and after 6 months of ETI treamtment (WP1), or probiotic/placebo (WP2. Levels of calprotectin, neopterin and myeloperoxidase will be measured.

CONTACTS AND LOCATIONS:
Locations (1):
- Oslo University Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No